CLINICAL TRIAL: NCT03851783
Title: Effect of Solar Powered Oxygen Delivery on Childhood Mortality in Uganda: A Cluster-Randomized Trial
Brief Title: Solar Oxygen Study
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Global Health Uganda LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084784
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Pneumonia; Hypoxemia
Keywords: solar; oxygen
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solar-powered oxygen (Experimental): Solar panels used to drive an oxygen concentrator will deliver medical grade oxygen at a rate of 1-5L/min, for the treatment of children with hypoxemia.
  Interventions: Device: Solar-powered oxygen
- Standard of care (No Intervention): Patients presenting with hypoxemia and pneumonia will be treated by standard of care prior to the implementation of solar-powered oxygen at a chosen site. This may include some allocation of oxygen via cylinders, but will likely be minimal or not available.

INTERVENTIONS:
Device: Solar-powered oxygen — Constant and reliable administration of oxygen, using solar panels to power an oxygen concentrator and deliver medical grade oxygen at 1-5L/min.
  Arms: Solar-powered oxygen

SUMMARY:
Globally, approximately 7.7 million children per year die before the age of 5 years. Infectious diseases account for a large proportion of these deaths, with pneumonia being the leading cause of mortality (2.1 million deaths/year). Most deaths occur in resource-poor settings in Asia and Africa. Oxygen (O2) therapy is essential to support life in these patients. Large gaps remain in the case management of children presenting to African hospitals with respiratory distress, including essential supportive therapies such as supplemental oxygen. In resource-constrained settings, oxygen delivery systems can lead to measurable improvements in survival from childhood pneumonia. A multihospital effectiveness study in Papua New Guinea demonstrated a reduction in mortality from childhood pneumonia from 5.0% to 3.2% (35% reduction in mortality) after implementation of enhanced oxygen delivery system. The investigators propose to investigate a novel strategy for oxygen delivery that could be implemented in remote locations with minimal access to an electrical power supply: solar-powered oxygen (SPO2).

DETAILED DESCRIPTION:
Clinical features of pneumonia in children include fever, respiratory distress, and hypoxemia. Respiratory distress is a useful clinical summary description with good inter-observer consistency among experienced medical practitioners. The following clinical signs may indicate increased work of breathing: sustained nasal flaring; indrawing (recession) of the bony structures of the chest wall (subcostal, intercostal, supraclavicular) on inspiration; tracheal tug; and deep breathing (acidotic or Kussmaul breathing). Respiratory distress is a sign that one or more serious pathological processes are at play: metabolic acidosis, fluid overload, acute lung injury, and/or co-morbid pneumonitis. Respiratory distress, together with alteration of consciousness, is a strong predictor of mortality in children with severe febrile illness in sub-Saharan Africa. The grim prognostic significance of respiratory distress applies to several disease states, irrespective of microbial etiology, including malaria as well as non-malaria febrile illness.

Arterial hypoxemia in pneumonia results from several mechanisms: pulmonary arterial blood flow to consolidated lung resulting in an intrapulmonary shunt, intrapulmonary oxygen consumption, and ventilation-perfusion mismatch. Hypoxemia is a risk factor for mortality in pediatric pneumonia, and was associated with a 5-fold increased risk of death in studies from Kenya and Gambia. In one report from Nepal, the prevalence of hypoxemia (SpO2 < 90%) in 150 children with pneumonia was 39% overall, with increasing rates of hypoxemia across strata of pneumonia severity (100% of very severe, 80% of severe and 17% of pneumonia patients). General features of respiratory distress were associated with hypoxemia in this study, including chest indrawing, lethargy, grunting, nasal flaring, cyanosis, inability to breastfeed or drink.

Oxygen is a lifesaving therapy for children with pneumonia and hypoxemia; however, challenges remain in oxygen delivery globally. Two main systems of oxygen delivery have been implemented and evaluated in resource-constrained settings, oxygen cylinders and oxygen concentrators. Oxygen cylinders are ready to use, simple to operate and do not require any electricity. However, cylinders are very costly and distribution and use is challenging. Oxygen concentrators have proven to be an effective means of delivering oxygen and are significantly less expensive that cylinders. However, oxygen concentrators require continuous and reliable electricity to operate which is not readily available in many regions, particularly in resource-limited settings where the majority of pneumonia deaths occur. In order to meet the demand for oxygen therapy in resource-limited settings, the investigators developed a novel strategy for oxygen delivery: solar-powered oxygen (SPO2). This system uses free inputs (sun and air) and could be implemented in remote locations with minimal access to an electrical power supply. Our group is the first to conduct rigorous scientific trials of SPO2.

To date, the investigators have accumulated substantial clinical experience with SPO2, having treated >150 hypoxemic children, over several years, at two Ugandan hospitals. Compared to other oxygen delivery methods, SPO2 is superior. SPO2 is more reliable than oxygen concentrators connected to grid electricity, because it is not affected by frequent power outages. SPO2 utilizes a renewable, sustainable and freely available source of energy. SPO2 is more reliable than compressed oxygen cylinders, which are frequently out of stock in the public hospital system. SPO2 is more user-friendly and safer for nurses than cylinders, which require physical strength to change regulators on high-pressure cylinders. SPO2 is less wasteful than cylinders, which tend to leak through ill-fitting regulators under real-world conditions.

The study is a multi-centre prospective evaluation of SPO2. The investigators will use a stepped-wedge cluster-randomized design to allow for robust scientific conclusions about the efficacy of SPO2. Importantly, demonstration of a mortality benefit of SPO2 will provide strong supportive evidence and could catalyse the widespread implementation of SPO2 in resource-limited settings across Africa and Asia.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 5 years
2. Hypoxemia (SpO2<92%) based on non-invasive pulse oximetry
3. Hospital admission warranted based on clinician judgment

Exclusion Criteria:

1. SpO2 ≥92%
2. Outpatient management
3. Denial of consent to participate in study

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2405 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Mortality | 48 hours
  Mortality at 48 hours after admission

SECONDARY OUTCOMES:
In hospital mortality | Until end of hospitalization (usually 3 to 7 days)
  Mortality during any point of hospital admission
Length of hospital stay | Until end of hospitalization (usually 3 to 7 days)
  Total length of hospital admission
Oxygen saturation | Until end of hospitalization (usually 3 to 7 days)
  Measured oxygen saturations before and after administration of oxygen, using standard procedures
Oxygen delivery system failure | Until end of trial (24 months)
  Number and duration of failures in any component of the oxygen delivery system, including solar panels, batteries, oxygen concentrator, and electrical components
Total costs of implementing solar-powered oxygen delivery systems | Until end of trial (24 months)
  Total costs of implementing solar-powered oxygen delivery systems at twenty sites, including installation, servicing and maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Hawkes, MD, PhD, Principal Investigator — University of Alberta; Robert O Opoka, MBChB, MPH, Principal Investigator — Makerere University/Global Health Uganda
Locations (20):
- Uganda (20):
  - Adumi Health Centre IV, Adumi
  - Apac District Hospital, Apac
  - Atiak Health Centre IV, Atiak
  - Bugobero Health Centre IV, Bugobero
  - Bukedea Health Centre IV, Bukedea
  - Bumanya Health Centre IV, Bumanya
  - Bundibugyo Hospital, Bundibugyo
  - Kagadi Hospital, Kagadi
  - Kalisizo Hospital, Kalisizo
  - Kamuli General Hospital, Kamuli
  - Kayunga District Hospital, Kayunga
  - Kidera Health Centre IV, Kidera
  - Kitagata Hospital, Kitagata
  - Kitgum General Hospital, Kitgum
  - Kyenjojo General Hospital, Kyenjojo
  - Lalogi Health Centre IV, Lalogi
  - Lyantonde Hospital, Lyantonde
  - Gombe Hospital, Mpigi
  - Muyembe Health Centre IV, Muyembe
  - Sembabule Health Centre IV, Sembabule

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turnbull H, Conroy A, Opoka RO, Namasopo S, Kain KC, Hawkes M. Solar-powered oxygen delivery: proof of concept. Int J Tuberc Lung Dis. 2016 May;20(5):696-703. doi: 10.5588/ijtld.15.0796. PMID 27084827
- [Background] Hawkes MT, Conroy AL, Namasopo S, Bhargava R, Kain KC, Mian Q, Opoka RO. Solar-Powered Oxygen Delivery in Low-Resource Settings: A Randomized Clinical Noninferiority Trial. JAMA Pediatr. 2018 Jul 1;172(7):694-696. doi: 10.1001/jamapediatrics.2018.0228. PMID 29800014
- [Derived] Conradi N, Opoka RO, Mian Q, Conroy AL, Hermann LL, Charles O, Amone J, Nabwire J, Lee BE, Saleh A, Mandhane P, Namasopo S, Hawkes MT. Solar-powered O2 delivery for the treatment of children with hypoxaemia in Uganda: a stepped-wedge, cluster randomised controlled trial. Lancet. 2024 Feb 24;403(10428):756-765. doi: 10.1016/S0140-6736(23)02502-3. Epub 2024 Feb 14. PMID 38367643
- [Derived] Conradi N, Mian Q, Namasopo S, Conroy AL, Hermann LL, Olaro C, Amone J, Opoka RO, Hawkes MT. Solar-powered oxygen delivery for the treatment of children with hypoxemia: protocol for a cluster-randomized stepped-wedge controlled trial in Uganda. Trials. 2019 Dec 5;20(1):679. doi: 10.1186/s13063-019-3752-2. PMID 31805985